CLINICAL TRIAL: NCT02713399
Title: High-resolution Imaging of Tear Film Thickness in Contact Lenses Wearers With Optical Coherence Tomography (OCT). A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Other Study IDs: OPHT-150116
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Contact Lens; Tear Film Thickness
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Soft Contact Lenses: healthy subjects wearing soft contact lenses
  Interventions: Device: Optical Coherence Tomography
- Rigid Contact Lenses: healthy subjects wearing rigid contact lenses
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography

SUMMARY:
A refractive error is the most common reason for reduced visual acuity. Myopia, hyperopia, astigmatism and presbyopia belong to the four basic refractive errors and, unfortunately, cannot be prevented. There are different tools to correct them, like spectacles, contact lenses, and refractive surgery. Many different contact lenses are available, the two large groups create rigid contact lenses and soft contact lenses. It is a common knowledge that the presence of a contact lens in the eye divides the tear film into the prelens and postlens tear film layers. In the present study we want to investigate the variability and reproducibility of prelens and postlens tear film thickness measurements.

ELIGIBILITY:
Inclusion criteria

* Men and women aged over 18 years
* Soft or rigid contact lenses wearers
* Schirmer Test ≥ 10 mm/5 min
* Tear Breakup Time (TBUT) ≥10 seconds

Exclusion Criteria:

* Participation in a clinical trial in the previous 3 weeks
* Presence of any abnormalities preventing reliable measurements as judged by the investigator
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 soft contact lens wearers 15 rigid contact lens wearers
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-03-16 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Pre lens and post lens tear film thickness | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria